CLINICAL TRIAL: NCT02670109
Title: High-dose Chemotherapy With Autologous Hematopoietic Stem Cell Transplantation as Adjuvant Treatment for Triple Negative Breast Cancer Patients Without Complete Pathological Response to Neoadjuvant Chemotherapy
Brief Title: Autologous Hematopoietic Stem Cell Transplantation as Adjuvant Treatment for Triple Negative Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCMNSZ REF 1239
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Triple-Negative Invasive Breast Carcinoma; Residual Tumor
MeSH Terms: conditions — Neoplasm, Residual | interventions — Carmustine; Cyclophosphamide; Carboplatin; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unique (Experimental): Patients will receive a high dose chemotherapy regimen, consisting in the administration of three medications: Carmustine (BCNU) 300mg/m2 or Busulfan 16 mg/kg (according to availability), Cyclophosphamide 80mg/kg, and Carboplatin 1400/m2.
  Then they will undergo an Autologous Hematopoietic Stem Cell Transplantation.
  Interventions: Drug: Carmustine; Drug: Cyclophosphamide; Drug: Carboplatin; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Busulfan

INTERVENTIONS:
Drug: Carmustine — 300mg/m2, IV, in 3 hours, during day -4
  Other Names: BCNU
Drug: Cyclophosphamide — 80mg/kg, IV, in 2 hours, during two days -2, -3
  Other Names: Cytoxan
Drug: Carboplatin — 1400/m2, IV, in 1 hour, during day -3
  Other Names: Paraplatin
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Transfusion, in 3 hours, during day 0
  Other Names: Peripheral blood autologous HSCT
Drug: Busulfan — 16mg/kg, Oral, during day -4
  Other Names: Myleran

SUMMARY:
Triple-negative breast cancer (TNBC) refers to any breast cancer that does not express estrogen receptor (ER), progesterone receptor (PR) or Her2/neu. Its incidence is approximately 180,000 cases per year. TNBC are known to be more aggressive with poor prognosis specially when no pathologic complete response (pCR) is achieved after neoadjuvant chemotherapy, with a higher risk of recurrence and a poor survival once that recurrence occurs. On the other hand, there is not a specific adjuvant or neoadjuvant treatment for these patients. Since autologous hematopoietic stem cell transplantation (HSCT) allows the usage of higher doses of chemotherapy, which results in higher cellular destruction with a decrease of hematological toxicity, it is proposed that this procedure is able to improve prognosis in TNBC patients with no pathologic complete response after neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Triple-negative breast cancer (TNBC) accounts for approximately 15%-25% of all breast cancer cases. TNBC are usually high-grade tumors, presented among younger women, African American and Hispanic women have a higher risk; generally in advanced stages when diagnosed, with visceral recurrence (liver, lung, brain). Standard treatment is surgery with adjuvant chemotherapy and radiotherapy. As a variation, neoadjuvant chemotherapy is very frequently used for triple-negative breast cancers, however, there is a lack of specific agents for this subset of patients, and, pathologic complete response does correlate with overall survival. At the moment, no optimal chemotherapy exists for TNBC patients who do not achieve a pCR.

According to the German group, in the triple negative subset, 31% of patients with neoadjuvant chemotherapy achieved pathologic complete response (pCR), which correlates with progression free survival (HR 6.02 for those who do not achieve pCR), and an overall survival (HR 12.41 for those who do not achieve pCR).

The usage of high-dose chemotherapy with autologous HSCT, is one of the therapies that have been studied in the patients with localized breast cancer aiming to improve its outcome. Autologous HSCT allows higher chemotherapy doses, which results in higher tumor cells destruction. Since 1980, several phase II studies were performed with high-dose chemotherapy and autologous HSCT, with an apparently initial benefit, thus this strategy was widely used outside controlled clinical trials. Afterward, the randomized studies did not show benefit in overall survival, causing this strategy to be abandoned.

It is important to highlight studies heterogeneity by means of different treatment options in both experimental and control group, besides, advances in autologous HSCT has significantly reduced the complexity, mobility, and mortality related to the chemotherapy treatment.

Two published studies including patients with localized TNBC, showed benefit in the progression free survival in the high-dose chemotherapy group, with a tendency to improved overall survival. One of them was performed by a german group, including patients with at least 9 positive nodes, which were randomized to receive two cycles of conventional dose chemotherapy followed by two cycles of high-dose chemotherapy with autologous HSCT versus four cycles of conventional dose chemotherapy followed by three cycles of dense dose chemotherapy, with granulocyte colony-stimulating factor (G-CSF) administration. Progression free survival was 76 months in the group of high dose chemotherapy versus 40.6 months in the conventional chemotherapy group, with an overall survival of 60 versus 44%, being statistically significant.

Our hypothesis is that patients with TNBC with a high risk of recurrence (no pCR) who undergo high-dose chemotherapy followed by autologous HSCT will have a higher overall survival compared to those who do not undergo the above mentioned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Triple Negative Breast Cancer diagnosis (no expression of hormonal receptors or Her2/neu)
* Previous administration of neoadjuvant chemotherapy (60 days maximum)
* No evidence of metastatic disease at inclusion
* Residual tumor in the breast and/or lymph nodes
* Normal renal, liver, heart, lung, and hematopoietic function

Exclusion Criteria:

* Pregnancy
* Disease progression during neoadjuvant therapy
* Other tumors
* Non triple negative breast cancer diagnosis
* Pathological Complete Response achieved

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | One year
  Time from diagnosis to death from any cause.

SECONDARY OUTCOMES:
Disease Free Survival | One year
  Time from ending primary treatment to relapse of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Eucario Leon Rodriguez, M.D., Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Monica M Rivera Franco, M.D.,MSc, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No